CLINICAL TRIAL: NCT02515578
Title: Southwest Health Extension Partnership to Enhance Research Dissemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-0403
Record Dates: First submitted 2015-07-15; First posted 2015-08-05 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Diseases
Keywords: Primary Health Care; Cardiovascular Diseases; Quality Improvement
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard practice transformation support (Active Comparator): Primary care practices will receive a cardiovascular care toolkit, practice facilitation, practice assessment with feedback, health information technology assistance, academic detailing, and periodic collaborative learning sessions
  Interventions: Other: Standard practice transformation support
- Enhanced practice transformation support (Experimental): Primary care practices will receive practice facilitation, practice assessment with feedback, health information technology assistance, academic detailing, and periodic collaborative learning sessions PLUS patient advisory council support and a modified cardiovascular care toolkit based on combined practice and patient input regarding the local context.
  Interventions: Other: Enhanced practice transformation support

INTERVENTIONS:
Other: Enhanced practice transformation support
  Arms: Enhanced practice transformation support
Other: Standard practice transformation support
  Arms: Standard practice transformation support

SUMMARY:
Heart disease and strokes cause one in three deaths reported each year in the United States. Primary care practices need to implement new research findings that help decrease patients' risk for heart disease and stroke. This project will help to build primary care practice capacity for quality improvement and change management in small and medium size primary care practices in Colorado and New Mexico. This project will also help practices implement patient-centered outcomes research findings.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) causes one in three deaths reported each year in the United States. Strategies derived from patient-centered outcomes research (PCOR) that address CVD risk factors can greatly reduce the burden of CVD. Primary care practices must transform to deliver a higher level of PCOR evidence-based prevention to decrease cardiovascular risk. PCOR interventions that emphasize patient-centered care including self-management support, team-based care, improved information systems, and active quality improvement have been shown to be effective. Practices often require assistance integrating new programs into clinical operations. Practice facilitation has been shown to enhance implementation of new programs for patients with chronic disease in primary care. Other methods of practice support, including academic detailing, collaborative learning sessions, and health information technology assistance, have also been shown to be effective, by themselves and in combination with practice facilitation. Patient involvement may also aid practice transformation. Increasingly, practices are actively including patients as part of the change process through the creation of patient advisory councils and including patients in practice quality improvement teams. Another method of patient involvement to inform implementation of evidence-based care is the Boot Camp Translation process, in which patients collaborate with primary care clinicians, staff members, and community members to translate best practices into culturally and community relevant implementation at the local level. However, while these efforts have had considerable success, no study has looked at the incremental value of adding patient engagement strategies to the more standard approaches to practice transformation listed above. This project would implement the Southwest Health Extension Program to Enhance Research Dissemination (SHEPERD) as a cooperative program to build primary care practice capacity for quality improvement, change management, and implementation of PCOR findings in small and medium size primary care practices in Colorado and New Mexico, with an initial focus on cardiovascular care. It also would conduct a cluster randomized trial with an external matched cohort control group to examine the Reach, Effectiveness, Adoption, Implementation, and Maintenance of two approaches to practice transformation to implement PCOR interventions for reducing cardiovascular risks in primary care practices, comparing the impact of 1) a standard practice transformation support intervention (including practice facilitation, practice assessment with feedback, HIT assistance, academic detailing, and collaborative learning sessions) to 2) an approach that adds patient engagement activities (including patient advisory councils and boot camp translation) as part of the practice transformation support. This project will provide critical information regarding the added value of patient engagement in practice transformation efforts and will also result in a network of practices across the region with increased capacity for practice transformation and implementation of PCOR findings.

ELIGIBILITY:
Inclusion Criteria:

* Must be staff or clinicians (including physicians, nurse practitioners, and physician assistants) in an enrolled primary care practice
* Primary care practices must be family medicine or general internal medicine practices with a maximum of ten lead clinicians
* Primary care practices must be either independent or, if part of a larger organization, demonstrate on careful screening that they do not receive significant quality improvement support from the larger organization

Exclusion Criteria:

* Primary care practices with more than 10 lead clinicians
* Non-independent primary care practices that receive significant quality improvement support from their system or organization
* Clinicians and staff who do not speak or read English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5508 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change of documentation of aspirin therapy in patients with ischemic vascular disease. | Baseline, 3, 6, 9, 12, and 15 months from baseline
  The percent of patients aged 18 years and older with Ischemic Vascular Disease (IVD) with documented use of aspirin or other antithrombotic. This is a practice-level indicator of documentation of care processes for cardiovascular disease.
Change of documentation of blood pressure in patients with a diagnosis of hypertension. | Baseline, 3, 6, 9, 12, and 15 months from baseline
  The percent of patients aged 18 - 85 who had a diagnosis of hypertension (HTN) and whose blood pressure (BP) was adequately controlled (<140/90) during the measurement year. This is a practice-level indicator of documentation of care processes for cardiovascular disease.
Change of documentation of blood pressure in patients with adequately controlled blood pressure. | Baseline, 3, 6, 9, 12, and 15 months from baseline
  The percent of patients aged 18 - 85 who had a diagnosis of hypertension (HTN) and whose blood pressure (BP) was adequately controlled (age 18-59 and/or people with diabetes or chronic kidney disease <140/90; age 60-85 <150/90) during the measurement year. This is a practice-level indicator of documentation of care processes for cardiovascular disease.
Change of documentation of fasting LDL in patients with a fasting LDL at or below the LDL goal. | Baseline, 3, 6, 9, 12, and 15 months from baseline
  The percent of patients aged 20 - 79 who had a fasting LDL test performed and whose risk-stratified fasting LDL is at or below the recommended LDL goal. This is a practice-level indicator of documentation of care processes for cardiovascular disease.
Change of documentation of patients who had a fasting LDL test performed and prescribed a statin based on risk. | Baseline, 3, 6, 9, 12, and 15 months from baseline
  The percent of patients aged 20 - 79 who had a fasting LDL test performed and who are prescribed a recommended dose of statin based on risk status if indicated. This is a practice-level indicator of documentation of care processes for cardiovascular disease.
Change of documentation of patients screened about tobacco use. | Baseline, 3, 6, 9, 12, and 15 months from baseline
  The percent of patients aged 18 years or older screened about tobacco use one or more times within 24 months AND who received cessation counseling intervention if identified as a tobacco user. This is a practice-level indicator of documentation of care processes for cardiovascular disease.

SECONDARY OUTCOMES:
Change of the documentation in primary care practice's. | Baseline, 9 and 15 months from baseline
  This primary care practice capacity to implement PCOR findings and improve quality and implementation of the planned comprehensive approach. The measure is based on practice-level scores of change process capacity, adaptive reserve, clinician experience and implementation of patient-centered medical home components.

CONTACTS AND LOCATIONS:
Overall Officials: W. Perry Dickinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Denver, Colorado, United States

REFERENCES:
- [Derived] Zittleman L, Westfall JM, Callen D, Herrick AM, Nkouaga C, Simpson M, Dickinson LM, Fernald D, Kaufman A, English AF, Dickinson WP, Nease DE Jr. Does engagement matter? The impact of patient and community engagement on implementation of cardiovascular health materials in primary care settings. BMC Prim Care. 2024 Apr 25;25(1):135. doi: 10.1186/s12875-024-02365-w. PMID 38664665
- [Derived] Fernald DH, Mullen R, Hall T, Bienstock A, Kirchner S, Knierim K, de la Cerda D, Callan D, Rhyne RL, Dickinson LM, Dickinson WP. Exemplary Practices in Cardiovascular Care: Results on Clinical Quality Measures from the EvidenceNOW Southwest Cooperative. J Gen Intern Med. 2020 Nov;35(11):3197-3204. doi: 10.1007/s11606-020-06094-5. Epub 2020 Aug 17. PMID 32808208
- [Derived] English AF, Dickinson LM, Zittleman L, Nease DE Jr, Herrick A, Westfall JM, Simpson MJ, Fernald DH, Rhyne RL, Dickinson WP. A Community Engagement Method to Design Patient Engagement Materials for Cardiovascular Health. Ann Fam Med. 2018 Apr;16(Suppl 1):S58-S64. doi: 10.1370/afm.2173. PMID 29632227